CLINICAL TRIAL: NCT05352334
Title: Comparison of High Intensity Interval Training Verses Aerobic Exercises on Emotional Intelligence of University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/516
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: High Intensity Interval Training; Aerobic Exercise

STUDY DESIGN:
Intervention Model Description: The participants fulfilling the inclusion criteria will be selected from above mentioned different government and private universities. The total number of participants in data collection procedure will be 44. Informed consent will be taken from all the students and self-administered questionnaire will be distributed to students for data collection procedure. The emotional intelligence and physical activity will be measured and collected through Schutte self-report Emotional Intelligence test (SSCEIT) and international physical activity questionnaire. The questionnaires for physical activity will consist of 12 questions and for SSCEIT consist of 33 questions. Emotional intelligence will be measured by schutte self-report emotional intelligence scale and physical activity will be measured by international physical activity questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental)
  Interventions: Diagnostic Test: self-report Emotional Intelligence test (SSCEIT)
- Aerobic Exercise (Experimental)
  Interventions: Diagnostic Test: self-report Emotional Intelligence test (SSCEIT)

INTERVENTIONS:
Diagnostic Test: self-report Emotional Intelligence test (SSCEIT) — The participants fulfilling the inclusion criteria will be selected from above mentioned different government and private universities. The total number of participants in data collection procedure will be 44. Informed consent will be taken from all the students and self-administered questionnaire will be distributed to students for data collection procedure. The emotional intelligence and physical activity will be measured and collected through Schutte self-report Emotional Intelligence test (SSCEIT) and international physical activity questionnaire. The questionnaires for physical activity will consist of 12 questions and for SSCEIT consist of 33 questions. Emotional intelligence will be measured by schutte self-report emotional intelligence scale and physical activity will be measured by international physical activity questionnaire.

SUMMARY:
High Intensity Interval Training verses Aerobic Exercises on Emotional Intelligence of University Students

DETAILED DESCRIPTION:
Null hypothesis: There is no difference in effects of high intensity interval training verses aerobic exercises on emotional intelligence of university students. Alternative hypothesis: there is difference in high intensity interval training and aerobic exercises on emotional intelligence of university students.

ELIGIBILITY:
Inclusion Criteria:

20-30 years old Both males & females Previously involved in any physical activity will be included in this study.

Exclusion Criteria:

Insomnia, ADHD, schizophrenia, bipolar disorder& depression, anxiety etc. Headache, epilepsy and seizures, stroke, Alzheimer disease , dementia & Parkinson's disease Drugs & alcohol abuse Any other known medical condition

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of High Intensity Interval Training verses Aerobic Exercises on Emotional Intelligence of University Students | 6 Months
  The main goal of this study is to determine the comparison of high intensity interval training and aerobic exercises on emotional intelligence. Physical activity (PA) is linked to emotional, physical, and social well-being. In terms of mental health, past research has revealed that people who participate in physical activity have higher psychological wellness and experience less stress and depression. Adolescents, undergraduate students, and the elderly were all involved in these results. Physical activity levels, on the other hand, are low in the university population over the world. According to a meta-analysis of college student physical activity practices, 40 to 50 percent do not satisfy the physical activity standards.

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided